CLINICAL TRIAL: NCT01849744
Title: A Phase I Study of VS-4718, a Focal Adhesion Kinase Inhibitor, in Subjects With Metastatic Non-Hematologic Malignancies
Brief Title: Phase I Dose Escalation Study of VS-4718 in Subjects With Metastatic Non-Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision to deprioritize the program.
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-4718-101
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Non Hematologic Cancers; Metastatic Cancer
Keywords: Focal Adhesion Kinase inhibitor; FAK inhibitor; Cancer Stem Cells; CSC
MeSH Terms: conditions — Neoplasm Metastasis | interventions — PND 1186

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VS-4718 (Experimental): Oral VS-4718 administered BID (QD during first cohort) during a 28 day cycle.
  Interventions: Drug: VS-4718

INTERVENTIONS:
Drug: VS-4718

SUMMARY:
This is a Phase I, open-label, multicenter, dose-escalation trial of VS-4718, a focal adhesion kinase inhibitor, in subjects with metastatic non-hematologic malignancies. This clinical study is comprised of 2 parts: Part 1 (Dose Escalation) and Part 2 (Expansion). The purpose of this study is to evaluate the safety (including the recommended Phase II dose), pharmacokinetics (the amount of VS-4718 in your blood) and the anti-cancer activity of VS-4718. The pharmacodynamic effects (genes or proteins that may predict or show how your body may respond to VS-4718) will also be examined in tumor biopsies and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histopathologically confirmed diagnosis of a metastatic non-hematologic malignancy.
* ECOG (Eastern Cooperative Oncology Group) performance status of ≤ 2
* Adequate renal function
* Adequate hepatic function (total bilirubin ≤ 1.5x ULN (upper limit of normal) for the institution; AST [aspartate transaminase] and ALT [alanine transaminase] ≤ 3x ULN, or ≤ 5x ULN if due to liver involvement by tumor).
* Adequate bone marrow function (hemoglobin ≥ 9.0 g/dL; unsupported platelets ≥ 100 x10 9 cells/L; absolute neutrophil count ≥ 1.5x10 9 cells/L
* Corrected QT interval (QTc) < 470 ms
* Subjects must have at least one tumor lesion that is suitable for repeat biopsy, and must agree to two tumor biopsies (pre- and post- treatment).
* Willing and able to participate in the trial and comply with all trial requirements.

Exclusion Criteria:

* Gastrointestinal (GI) condition which could interfere with the swallowing or absorption of study medication.
* Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases).
* History of upper gastrointestinal bleeding, ulceration, or perforation within 12 months.
* Known history of stroke or cerebrovascular accident within 6 months.
* Subjects being actively treated for a secondary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of VS-4718 in subjects with metastatic non-hematologic malignancies | Expected average of 12 weeks from start of treatment to end of treatment
  Serious Adverse events, Adverse events and their frequency, duration and severity, physical examination, laboratory parameters, vital signs and ECGs as determined based on CTCAE (Common Toxicity Criteria for Adverse Effects) V4.03. A Safety monitoring committee will review safety information.
Establish the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of VS-4718 in subjects with metastatic non-hematologic malignancies | From start of treatment to end of cycle 1 (4 week cycles)
  The RP2D will be determined based on the maximum tolerated dose (MTD) of VS-4718 as determined by number of participants with dose limiting toxicities related to VS-4718. Observations related to pharmacokinetics, pharmacodynamics, and any VS-4718 related toxicities may be included in the rationale supporting the RP2D and will not exceed the MTD.

SECONDARY OUTCOMES:
Evaluate the efficacy of VS-4718 | Every 8 weeks to end of treatment, expected average of 16 weeks
  Response rate and progression-free survival as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1
Evaluate duration of response to VS-4718 compared with duration of response to prior therapy. | Expected average of 16 weeks from start of treatment to end of treatment
Assess the pharmacokinetics of VS-4718 | Time points on Day 1, 2, 8, 15, 16, and 29
  PK (pharmacokinetics) parameters, including but not limited to clearance, plasma concentration, AUC (Area Under Curve, 0-24 and 0-t), Cmax, Tmax, and T1/2
Evaluate biomarkers of VS-4718 activity | Day 1 and Day 15 of treatment
  Pre and post dose biomarker analysis in serum and tumor samples to identify possible prognostic factors to VS-4718 response
Examine if the tumor expression status of pFAK and other plasma biomarkers correlates with response to VS-4718 therapy | From start of treatment to end of treatment, an expected average of 16 weeks
  Tumor expression status (pFAK, cancer stem cells, CSC, and other biomarkers) compared with response to VS-4718, as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Samuel Oschin Comprehensive Cancer Institute, Cedars-Sinai Medical Center, Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Washington University School of Medicine, Division of Oncology, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee